CLINICAL TRIAL: NCT00509639
Title: Phase III Study to Evaluate the Effect of 10% Metronidazole Ointment, Applied Topically Three Times a Day in and Around the Anus and the Change in Perianal Crohn's Disease Activity
Brief Title: Evaluation of Topical 10% Metronidazole Ointment for the Treatment of Active Perianal Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MET/01
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole 10% ointment (Experimental): Metronidazole 10% ointment
  Interventions: Drug: 10% Metronidazole Ointment
- Placebo ointment (Placebo Comparator): Placebo ointment
  Interventions: Drug: 10% Metronidazole Ointment

INTERVENTIONS:
Drug: 10% Metronidazole Ointment — Metronidazole 10% ointment applied perianally three times daily for four weeks. Placebo ointment applied perianally three times daily for four weeks

SUMMARY:
The purpose of this study is to compare changes in Perianal Crohn's Disease following use of locally applied 10% metronidazole ointment and a placebo.

DETAILED DESCRIPTION:
Anorectal Crohn's disease is one of the most problematic and debilitating conditions encountered in colorectal practise. The condition is usually chronic, debilitating, and frequently refractory to current medications. Failure to respond to medical therapy may ultimately result in proctocolectomy and ileostomy, even in the absence of more proximal colonic disease. Isolated anorectal Crohn's disease is reported in 3 to 5% of Crohn's patients. In Crohn's patients as a whole, anorectal involvement is reported in up to one third to one half of patients, in addition to either colonic or enteric Crohn's disease. In spite of the previously reported painless nature of anorectal Crohn's disease, it is the author's experience that the condition can be inordinately painful due to deeply eroding fissures, oedematous skin tags, and painful induration of the perianal region.

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease (diagnosed by radiology, endoscopy and pathology), with anorectal involvement.
* Have had perianal symptoms for longer than 3 months
* Have a PCDAI of 5 or above at baseline
* Subjects can be on concomitant medication. Acceptable regimes are:-
* Aminosalicylates at a dosage that has been stable for more than 4 weeks before screening;
* Oral corticosteroids <40mg per day that has been stable for more than 3 weeks;
* Methotrexate given for at least 3 months that has been stable for more than 4 weeks; Azathioprine or mercaptopurine given for at least 6 months at dosage that has been stable for more than 8 weeks;
* Antibiotics at a dosage that has been stable for 4 weeks (subjects may be on oral metronidazole but on a dose not more than 750mg per day),
* Cycolsporin for more than 3 months and on a stable dose for more than 4 weeks;
* Patients who have been treated with Infliximab must have received their initial dose 3 months before starting study medication and their most recent dose at least 8 weeks before starting study medication and not receive an infusion whilst in the double-blind treatment phase of the study for 4 weeks. During the second 4 week open stage of the study patients can commence again a maintenance regime with Infliximab treatment if deemed necessary
* Any patients not on concurrent medication must have been off medication for at least 4 weeks before screening.
* If patients have Setons these must have been in place for at least 4 weeks prior to screening.
* Subjects must be aged 18 years or over and of the legal age of consent.
* If female, the subject must not be lactating and must be (a) post- menopausal, (b) surgically sterilised, or (c) have a negative pregnancy test result prior to entry into the study and will use double- barrier methods of contraception (two separate methods of birthcontrol one of which may include oral contraception) for the duration of the study.
* Must have provided written informed consent to participate.

Exclusion Criteria:

* They have had surgery to the anus or rectum in the past 4 weeks;
* They have a perianal abscess requiring incision and drainage;
* They have a stoma of less than 6 months duration;
* Allergic to metronidazole;
* Are taking any prohibited medication.
* Deemed mentally incompetent.
* Considered by their physician unlikely to be able to comply with the protocol.
* Taken part in an experimental drug study in the preceding three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of 10% metronidazole ointment, applied topically three times a day, in and around the anus, on the change in perianal Crohn's disease activity. | Four weeks
  Perianal Crohn's Disease Activity Index

SECONDARY OUTCOMES:
To evaluate and compare the relief of perianal pain and discomfort associated with Crohn's disease, against placebo. | 4 weeks
  Perianal Crohn's Disease Activity Index plus Visual Analogue Scale for perianal pain
To evaluate and compare Patient Global Impression of Improvement | 4 weeks
  Patient Global Impression of Improvement (numerical scale)
To compare visual improvement (using photographic documentation assessed by a blinded independent observer) | 4 weeks
  Photographic record
To compare Quality of Life assessments | 4 weeks
  Short Form 12 Questionnaire
To evaluate and compare the number of analgesics required prior to treatment and to that required by the treatment and placebo group | 4 weeks
  Usage of analgesics during the treatment period
To evaluate and compare fistula healing | 4 weeks
  Visual assessment of fistula healing

CONTACTS AND LOCATIONS:
Overall Officials: Emin Carapeti, BSc,MBBS,MD,, Principal Investigator — St Thomas Hospital, London
Locations (11):
- Washington University School of Medicine, St Louis, Missouri, United States
- United Kingdom (10):
  - Derby City General Hospital, Derby, Derbyshire
  - Leicester General Hospital, Leicester, Leicestershire
  - Monklands Hospital, Airdrie
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - University Hospital of Wales, Cardiff
  - University Hospital of Warwick and Coventry, Coventry
  - St Marks Hospital, Harrow
  - St Thomas Hospital, London
  - Peterborough District Hospital, Peterborough

REFERENCES:
- [Derived] Maeda Y, Ng SC, Durdey P, Burt C, Torkington J, Rao PK, Mayberry J, Moshkovska T, Stone CD, Carapeti E, Vaizey CJ; Topical Metronidazole in Perianal Crohn's Study Group. Randomized clinical trial of metronidazole ointment versus placebo in perianal Crohn's disease. Br J Surg. 2010 Sep;97(9):1340-7. doi: 10.1002/bjs.7121. PMID 20632322